CLINICAL TRIAL: NCT06492616
Title: Elacestrant Versus Standard Endocrine Therapy in Women and Men With Node-positive, Estrogen Receptor-positive, HER2-negative, Early Breast Cancer With High Risk of Recurrence-A Global, Multicenter, Randomized, Open-label Phase 3 Study
Brief Title: A Study of Elacestrant Versus Standard Endocrine Therapy in Women and Men With ER+,HER2-, Early Breast Cancer With High Risk of Recurrence
Acronym: ELEGANT
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Stemline Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STML-ELA-0422; 2024-515445-42-00 (EU CTIS Number)
Record Dates: First submitted 2024-07-01; First posted 2024-07-09 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Breast Cancer
Keywords: ELEGANT; Breast Cancer Stage II; Breast Cancer Stage III; Breast Cancer Female; Breast Cancer, Male; High-Risk Breast Cancer; High Risk Breast Carcinoma; ER-positive Breast Cancer; ER-positive HER-2 Negative Breast Cancer; ER Positive/HER2 Low Breast Cancer; Breast Cancer, ER+, HER2-; Adjuvant; Adjuvant Therapy
MeSH Terms: conditions — Breast Neoplasms; Breast Neoplasms, Male | interventions — elacestrant; Anastrozole; Letrozole; exemestane; Tamoxifen

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Elacestrant (Experimental): Participants will receive 345 milligrams (mg) elacestrant once daily (QD) for 5 years.
  Interventions: Drug: Elacestrant
- Standard of Care (SoC) Endocrine Therapy (Experimental): Participants will receive the SoC endocrine therapy that was used prior to randomization:
  * AI (anastrozole 1 mg QD, letrozole 2.5 mg QD, or exemestane 25 mg QD); or
  * Tamoxifen 20 mg QD
  Interventions: Drug: Anastrozole; Drug: Letrozole; Drug: Exemestane; Drug: Tamoxifen

INTERVENTIONS:
Drug: Elacestrant — Administered as oral tablets
  Arms: Elacestrant
Drug: Anastrozole — Administered as oral tablets
  Arms: Standard of Care (SoC) Endocrine Therapy
Drug: Letrozole — Administered as oral tablets
  Arms: Standard of Care (SoC) Endocrine Therapy
Drug: Exemestane — Administered as oral tablets
  Arms: Standard of Care (SoC) Endocrine Therapy
Drug: Tamoxifen — Administered as oral tablets
  Arms: Standard of Care (SoC) Endocrine Therapy

SUMMARY:
The primary goal of this study is to evaluate the effectiveness of elacestrant versus standard endocrine therapy in participants with node-positive, Estrogen Receptor-positive (ER+), Human Epidermal Growth Factor-2 negative (HER2-) early breast cancer with high risk of recurrence.

ELIGIBILITY:
Key Inclusion Criteria:

* Histopathologically or cytologically confirmed ER-positive (≥ 10% by immunohistochemistry [IHC]), HER2-negative [IHC = 0 or 1, or (IHC = 2 and in situ hybridization [ISH]-negative)] on tumor biopsy or final surgical pathology specimen early stage resected invasive breast cancer without evidence of recurrence or distant metastases, per local laboratory, according to the American Society of Clinical Oncology (ASCO)/College of American Pathologists (CAP) guidelines
* Participants considered at high risk of recurrence at initial staging
* Participants who have received at least 24 months but not more than 60 months of endocrine therapy (AIs or tamoxifen) with or without a CDK 4 and CKD 6 inhibitor (CDK4/6i)
* Participants who received prior CDK4/6i or a poly adenosine diphosphate-ribose polymerase (PARP) inhibitor must have already completed or discontinued these treatments.

Key Exclusion Criteria:

* Participants with inflammatory breast cancer
* History of any prior (ipsilateral and/or contralateral) invasive breast cancer
* Participant with history of malignancy within 3 years of the date of randomization, except for adequately treated basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix
* Participants who have had more than a 6-month continuous interruption of prior SoC adjuvant endocrine therapy or who discontinued adjuvant endocrine therapy more than 6 months prior to randomization

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4220 (Estimated)
Dates: Start 2024-09-27 (Actual); Primary Completion 2029-08 (Estimated); Study Completion 2032-10 (Estimated)

PRIMARY OUTCOMES:
Invasive Breast Cancer-Free Survival (IBCFS) | Up to 5 years
  Assessed by the time from date of randomization to the date of first occurrence of:
  * Ipsilateral invasive breast tumor recurrence
  * Local/regional invasive breast cancer recurrence
  * Distant recurrence
  * Contralateral invasive breast cancer, or
  * Death attributable to any cause

SECONDARY OUTCOMES:
Distant Relapse-Free Survival (DRFS) | Up to 5 years
  Assessed by the time from date of randomization to the date of first occurrence of:
  * Distant recurrence, or
  * Death attributable to any cause
Overall Survival (OS) | Up to 5 years
Invasive Disease-Free Survival (IDFS) | Up to 5 years
  Assessed by the time from date of randomization to the date of first occurrence of:
  * Local/regional recurrence
  * Contralateral recurrence
  * Second primary non-breast invasive cancer
  * Distant recurrence, or
  * Death attributable to any cause
Number of Participants With Adverse Events (AEs) | Up to 5 years plus 28 days
Change from Baseline in Global Health Status Quality of Life Scale score, as Assessed by the European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) | Baseline, Month 6, Annually at Years 1, 2, 3, 4, 5
Change from Baseline in the Physical Functioning Sub-Scale Score as Assessed by EORTC QLQ-C30 | Baseline, Month 6, Annually at Years 1, 2, 3, 4, 5
Change From Baseline in the Breast Cancer Endocrine Therapy Symptoms Sub-Scale Score, as Assessed by the EORTC Quality of Life Breast Cancer Questionnaire module (EORTC QLQ-BR42) | Baseline, Month 6, Annually at Years 1, 2, 3, 4, 5
Change From Baseline in Side Effects, as Assessed by the Question 168 of the European Organization for the Research and Treatment of Cancer Question Library (EORTC Q168) | Baseline, Month 6, Annually at Years 1, 2, 3, 4, 5
Area Under the Plasma Concentration Versus Time Curve at Steady State (AUCss) of Elacestrant | Predose up to 4 hours postdose
Maximum Plasma Concentration at Steady State (Cmaxss) of Elacestrant | Predose up to 4 hours postdose

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Stemline Therapeutics, Inc.
Locations (517):
- United States (153):
  - Southern Cancer Center, PC, Daphne, Alabama
  - Ironwood Cancer and Research Centers, Chandler, Arizona
  - Banner MD Anderson Cancer Center, Gilbert, Arizona
  - Mayo Clinic, Scottsdale, Arizona
  - Arizona Clinical Research Center, Inc., Tucson, Arizona
  - University of Arizona Cancer Center, Tucson, Arizona
  - Highlands Oncology Group, PA, Springdale, Arkansas
  - Comprehensive Blood & Cancer Center, Bakersfield, California
  - UCSF Cancer Center Berkeley, Berkeley, California
  - City of Hope National Medical Center, Duarte, California
  - UCSF Wash Cancer CNTR, Fremont, California
  - UC San Diego Moores Cancer Center, La Jolla, California
  - Helios Clinical Research, Long Beach, California
  - Cancer and Blood Research Center, LLC, Los Alamitos, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA Department of Medicine - Hematology/Oncology, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - UC Irvine Health, Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford Women's Cancer Center, Palo Alto, California
  - Dignity Health dba Health Research Institute, Sacramento, California
  - Sutter Institute for Medical Research, Sacramento, California
  - UCSF Zuckerberg SF General, San Francisco, California
  - University of California, San Francisco (UCSF), San Francisco, California
  - Southern California Kaiser Medical Center-San Marcos Medical, San Marcos, California
  - UCSF Cancer Center San Mateo, San Mateo, California
  - Sansum Clinic, Solvang, California
  - Torrance Memorial Physician Network- Cancer Care, Torrance, California
  - St.Joseph Hospital- Cancer Centers of Colorado, Denver, Colorado
  - Rocky Mountain Cancer Centers, LLP, Lone Tree, Colorado
  - AHMG Hematology and Oncology, Parker, Colorado
  - Cancer Care at CommonSpirit St. Anthony North Hospital, Westminster, Colorado
  - Yale New Haven Hospital- Yale Cancer Center, New Haven, Connecticut
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - The George Washington Medical Faculty Associates, Washington D.C., District of Columbia
  - Boca Raton Regional Hospital (BRRH) - Lynn Cancer Institute, Boca Raton, Florida
  - Florida Cancer Specialists, Fort Myers, Florida
  - Mayo Clinic, Jacksonville, Florida
  - Helios Clinical, Lakeland, Florida
  - Miami Cancer Institute at Baptist Health Inc., Miami, Florida
  - University of Miami, Miami, Florida
  - AdventHealth Orlando Infusion Center, Orlando, Florida
  - Cancer Care Centers of Brevard (CCCB) - Palm Bay, Palm Bay, Florida
  - Memorial Healthcare System, Pembroke Pines, Florida
  - Miami Cancer Institute at Plantation, Plantation, Florida
  - Florida Cancer Specialists, St. Petersburg, Florida
  - Comprehensive Hematology Oncology, St. Petersburg, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Florida Cancer Specialists, West Palm Beach, Florida
  - University Blood & Cancer Center, LLC, Athens, Georgia
  - Winship Cancer Institute, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Kaiser Permanente Hawaii Moanalua Medical Center, Honolulu, Hawaii
  - Illinois Cancer Specialists, Arlington Heights, Illinois
  - Northwestern Memorial Hospital, Chicago, Illinois
  - RUSH MD Anderson Cancer Center, Chicago, Illinois
  - Northwest Cancer Centers, PC, Dyer, Indiana
  - Mission Cancer and Blood, Des Moines, Iowa
  - Cancer Center of Kansas, Wichita, Kansas
  - University Medical Center-New Orleans, New Orleans, Louisiana
  - Mercy Medical Center, Baltimore, Maryland
  - Ascension St. Agnes Hospital, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Maryland Oncology Hematology, P.A., Columbia, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mass General North Shore Cancer Center, Danvers, Massachusetts
  - Dana Farber Cancer Institute at Foxborough, Foxborough, Massachusetts
  - Dana Farber Cancer Institute - Merrimack Valley, Methuen, Massachusetts
  - Dana-Farber Cancer Institute at Milford Regional, Milford, Massachusetts
  - Mass General Cancer Center at Newton-Wellesley Hospital's Vernon Cancer Center, Newton, Massachusetts
  - Dana-Farber/Brigham and Women's Cancer Center (DF/BWCC) in Clinical Affiliation with South Shore Hospital, South Weymouth, Massachusetts
  - Mass General - North Shore Cancer Center, Waltham, Massachusetts
  - The Cancer & Hematology Centers, Grand Rapids, Michigan
  - Mayo Clinic Health System - Albert Lea, Albert Lea, Minnesota
  - Mayo Clinic - Mankato, Mankato, Minnesota
  - Allina Health Cancer Institute - Abbott Northwestern Hospital, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Siteman Cancer Center, St Louis, Missouri
  - NHO Revive Research Institute LLC, Lincoln, Nebraska
  - Oncology Hematology West, PC dba Nebraska Cancer Specialists - Legacy, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - MD Anderson Cancer Center at Cooper, Camden, New Jersey
  - Summit Medical Group, Florham Park, New Jersey
  - John Theurer Ctr-Hackensack UMC, Hackensack, New Jersey
  - Rutgers Cancer Institute, New Brunswick, New Jersey
  - Exigent Research LLC/New Mexico Oncology Hematology Consultants Ltd., Albuquerque, New Mexico
  - Kings County Hospital Center, Brooklyn, New York
  - Hematology Oncology Associates of Central New York, PC, East Syracuse, New York
  - Cayuga Medical Center, Ithaca, New York
  - NYU Langone Hospital-Long Island, Mineola, New York
  - The Blavatnik Family - Chelsea Medical Center at Mount Sinai, New York, New York
  - Laura and Isaac Perlmutter Cancer Center/NYU Langone Health, New York, New York
  - Mount Sinai West, New York, New York
  - Icahn School of Medicine Mount Sinai, New York, New York
  - Columbia University Medical Center, New York, New York
  - University of Rochester Medical, Rochester, New York
  - Stony Brook University Cancer Center, Stony Brook, New York
  - Clinical Research Alliance, Inc., Westbury, New York
  - Duke Cancer Institute, Durham, North Carolina
  - Cape Fear Valley Medical Center, Fayetteville, North Carolina
  - Cone Health Cancer Center at Wesley Long, Greensboro, North Carolina
  - Miami Valley Hospital South, Centerville, Ohio
  - MetroHealth, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Oncology_Hematology Care Clinical Trials, LLC, Fairfield, Ohio
  - Oklahoma Cancer Specialists and Research Institute (OCSRI) - Tulsa Cancer Center, Tulsa, Oklahoma
  - Providence Cancer Institute Franz Clinic, Portland, Oregon
  - Oregon Oncology Specialists, Salem, Oregon
  - Northwest Cancer Specialists, P.C., Tigard, Oregon
  - Lehigh Valley Health Network - Cedar Crest, Allen, Pennsylvania
  - Consultants In Medical Oncology and Hematology, P.C., Broomall, Pennsylvania
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Holy Redeemer Hospital And Medical Center, Meadowbrook, Pennsylvania
  - Alliance Cancer Specialists, PC, Media, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - Cancer Care Associates of York, Inc., York, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Hollings Cancer Center, Charleston, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Baptist Cancer Center, Memphis, Tennessee
  - SCRI Oncology Partners, Nashville, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Henry - Joyce Cancer Clinic, Nashville, Tennessee
  - Hendrick Cancer Center, Abilene, Texas
  - Texas Oncology-Northeast Texas, Allen, Texas
  - Texas Oncology - DFW, Dallas, Texas
  - Oncology Consultants, P.A., Houston, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - O'Quinn Medical Tower - McNair Campus, Houston, Texas
  - Texas Oncology - San Antonio, New Braunfels, Texas
  - Texas Oncology-Gulf Coast, Pearland, Texas
  - Mays Cancer Center, San Antonio, Texas
  - Texas Oncology- Central South, Weslaco, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
  - University of Vermont Medical Center, Burlington, Vermont
  - Inova Schar Cancer Institute, Fairfax, Virginia
  - Virginia Oncology Associates, Newport News, Virginia
  - Virginia Cancer Institute, Richmond, Virginia
  - Oncology & Hematology Associates of Southwest Virginia, Inc, Wytheville, Virginia
  - Vista Oncology, Olympia, Washington
  - Virginia Mason Medical Center, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Fred Hutchinson Cancer Center, Seattle, Washington
  - Cancer Care Northwest, Spokane Valley, Washington
  - MultiCare Cancer Institute - Tacoma, Tacoma, Washington
  - Northwest Medical Specialties PLLC, Tacoma, Washington
  - Mayo Clinic Health System - Eau Claire, Eau Claire, Wisconsin
  - Mayo Clinic Health System - La Crosse, La Crosse, Wisconsin
  - University of Wisconsin Carbone Cancer Center- University Hospital, Madison, Wisconsin
  - UW Cancer Center at ProHealth Care, Waukesha, Wisconsin
- Argentina (11):
  - (COIBA)Centro de Oncologia e Investigacion Buenos Aires, Berazategui, Buenos Aires
  - Fundacion Respirar, Buenos Aires, Buenos Aires F.D.
  - Organizacion Medica de Investigacion (OMI), Buenos Aires, Buenos Aires F.D.
  - Centro de Investigación CIPREC, C.a.b.a., Buenos Aires F.D.
  - Centro Oncológico Korben, CABA, Buenos Aires F.D.
  - Centro Medico Privado CEMAIC, Córdoba, Córdoba Province
  - Inst Med Fund Estudios Clinicos, Rosario, Santa Fe Province
  - Instituto de Oncologia de Rosario, Rosario, Santa Fe Province
  - Clinica Adventista Belgrano, Buenos Aires, Tucumán Province
  - Instituto Argentino de Diagnostico y Tratamiento, Buenos Aires
  - Centro Oncologico de Excelencia, San Juan
- Australia (22):
  - St Vincent's Hospital Sydney, Darlinghurst, New South Wales
  - Lake Macquarie Private Hospital - Oncology, Gateshead, New South Wales
  - St George Hospital - Medical Oncology, Kogarah, New South Wales
  - Lismore Base Hospital - Cancer Care , Haematology Unit, Lismore, New South Wales
  - Macquarie University, Macquarie Park, New South Wales
  - Mater Hospital Sydney, North Sydney, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Icon Cancer Centre Townsville, Hyde Park, Queensland
  - Icon Cancer Centre Southport, Southport, Queensland
  - Icon Cancer Centre Wesley, Auchenflower, Quuensland
  - Cancer Research SA, Adelaide, South Australia
  - Royal Adelaide Hospital - Oncology, Adelaide, South Australia
  - Flinders Medical Centre, Bedford Park, South Australia
  - Icon Cancer Centre Kurralta Park, Kurralta Park, South Australia
  - The Queen Elizabeth Hospital, Woodville, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Medical Centre, Clayton, Victoria
  - Northern Hospital, Epping, Victoria
  - Goulburn Valley Health, Shepparton, Victoria
  - Breast Cancer Research Centre, Nedlands, Western Australia
  - Icon Cancer Centre Hobart, Hobart
  - Mid North Coast Cancer Institute, Port Macquarie
- Austria (5):
  - Universitätsklinikum Krems, Krems, Lower Austria
  - Universitatsklinikum St. Polten, Sankt Pölten, Lower Austria
  - LKH Hochsteiermark, Leoben, Styria
  - Brustgesundheitszentrum Süd, Weiz, Styria
  - Hanusch Krankenhaus, Vienna
- Belgium (12):
  - Algemeen Ziekenhuis Klina, Brasschaat, Antwerpen
  - Clnique Saint Pierre Ottignies - Oncologie-Hématologie, Ottignies, Brabant Wallon
  - Edith Cavell Inter-regional Hospital Centre (CHIREC) - Delta Hospital, Aalst, Brussels Capital
  - CHU Saint-Pierre, Brussels, Brussels Capital
  - Grand Hopital de Charleroi - Site Les Viviers, Charleroi, Hainaut
  - Jessa Ziekenhuis - Campus Virga Jesse - Medische Oncologie, Hasselt, Limburg
  - VITAZ Campus Sint-Niklaas Moerland, Sint-Niklaas, Oost-Vlaanderen
  - UZ Leuven, Leuven, Vlaams Brabant
  - Institut Jules Bordet, Brussels
  - CHU De Liège - Oncologie Médicale, Liège
  - CHC - Oncologie - Hémato-Immunopatho, Liège
  - CHU UCL Namur - Site Ste Elisabeth - Oncologie, Namur
- Brazil (29):
  - Instituto D'Or de Pesquisa e Ensino (Oncocentro Servicos Medicos e Hospitalares LTDA), Fortaleza, Ceará
  - Centro de Pesquisas Clínicas em Oncologia, Cachoeiro de Itapemirim, Espírito Santo
  - CEDOES - Centro de Pesquisa Clinica e Diagnostico do Espirito Santo LTDA, Vitória, Espírito Santo
  - Hospital Araujo Jorge, Goiânia, Goiás
  - CETUS Oncologia S.A, Belo Horizonte, Minas Gerais
  - Hospital Santa Cruz Sociedade Anonima, Curitiba, Paraná
  - Centro Integrado Oncologia Curitiba, Curitiba, Paraná
  - Instituto de Câncer de Londrina, Londrina, Paraná
  - CTO Centro de Tratamento Oncologico LTDA, Belém, Pará
  - Hospital da Fundacao Oswaldo Aranha, Volta Redonda, Rio de Janeiro
  - Sociedade Beneficência e Caridade de Lajeado (Hospital Bruno Born), Lajeado, Rio Grande do Sul
  - Futtura Oncologia, Porto Alegre, Rio Grande do Sul
  - Centro Gaucho Integrado de Oncologia, Hematologia, Ensino e Pesquisa - Hospital Mae de Deus, Porto Alegre, Rio Grande do Sul
  - Fundação PIO XII - Hospital de Amor Amazônia, Porto Velho, Rondônia
  - Centro de Pesquisas Oncologicas - CEPON, Florianópolis, Santa Catarina
  - Clinica de Neoplasias Litoral, Itajaí, Santa Catarina
  - Fundação Pio XII - Hospital de Amor de Barretos, Barretos, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo (ICESP), Barueri, São Paulo
  - Universidade de Sao Paulo (USP) - Hospital das Clinicas da Faculdade de Medicina de Ribeirao Preto (HCFMRP), Ribeirão Preto, São Paulo
  - Hospital de Base de São José do Rio Preto - CIP, São José do Rio Preto, São Paulo
  - Instituto Brasileiro de Controle do Cancer - ibcc - Hematology / Oncology, São Paulo, São Paulo
  - PUCRS - Hospital São Lucas, Porto Alegre
  - Instituto Nacional do Cancer - INCA-HC III, Rio de Janeiro
  - Instituto de Educacao, Pesquisa e Gestao em Saude, Rio de Janeiro
  - Clínica de Pesquisas e Centro de Estudos em Oncologia Ginecológica e Mamária Ltda, São Paulo
  - A.C.Camargo Cancer Center, São Paulo
  - Instituto de Assistencia Medica ao Servidor Publico Estadual (IAMSPE), São Paulo
  - Onco Star SP Oncologia LTDA (Onco Star), São Paulo
  - Hospital Universitario y Politecnico La Fe - Oncología Médica, Valência
- Canada (10):
  - BC Cancer -Surrey, Surrey, British Columbia
  - BC Cancer Agency, Vancouver, British Columbia
  - Royal Victoria Regional Health Centre; c/o Oncology Clinical Trials, Barrie, Ontario
  - London Health Sciences Centre, London, Ontario
  - St. Michaels Hospital, Toronto, Ontario
  - Mount Sinai Hospital - Study Supplies, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
  - Centre hospitalier régional de Lanaudière, Saint-Charles-Borromée, Quebec
  - Regional Hospital Saint-Jerome, Saint-Jérôme, Quebec
  - Hôpital du Saint-Sacrement, Québec
- Czechia (4):
  - Masarykuv onkologicky ustav - Klinika komplexni onkol. pece, Brno, Brno-město
  - Multiscan s.r.o., Hořovice, Stredoceský Kraj
  - FN Kralovske Vinohrady - Radioterapeuticka a onkologicka klinika, Prague
  - Fakultni Thomayerova nemocnice - Onkologicka klinika, Prague
- Denmark (3):
  - Hillerod Hospital, Hillerød, Capital
  - Odense Universitetshospital - Oncology, Odense, Region Syddanmark
  - Soenderborg Sygehus, Sønderborg, Region Syddanmark
- Finland (6):
  - Docrates Mehiläinen Syöpäsairaala, Mehiläinen Oy, Helsinki, Etelä-Suomen Lääni
  - Tampere University Hospital, Tampere, Etelä-Suomen Lääni
  - Turku University Hospital, Turku, Etelä-Suomen Lääni
  - Helsinki University Central Hospital (HUCH) - Meilahden Sair, Helsinki, Länsi-Suomen Lääni
  - Vaasa Central Hospital, Vaasa, Länsi-Suomen Lääni
  - Kuopio University Hospital, Pohjois-Savon hyvinvointialue, Kuopio, Northern Savonia
- France (22):
  - Centre Hospitalier Regional et Universitaire (CHRU) de Besancon - L'Hopital Jean Minjoz, Besançon, Alpes-Maritimes
  - Polyclinique Saint George, Nice, Alpes-Maritimes
  - Inst Cancerologie Strasbourg Europe, Strasbourg, Alsace
  - CHU de Grenoble, Grenoble, Auvergne-Rhône-Alpes
  - Centre de cancerologie Les Dentellieres, Valenciennes, Hauts-de-France
  - Ct Oncologie Radiotherapie CORT 37, Chambray-lès-Tours, Indre-et-Loire
  - Hopital Universitaire Dupuytren, Limoges, Limousin
  - Polyclinique de Blois, La Chaussée-Saint-Victor, Loir-et-Cher
  - Institut de Cancerologie de l'Ouest - Oncology, Saint-Herblain, Loire-Atlantique
  - ICONE, Bezannes, Marne
  - CRLCC Jean Godinot, Reims, Marne
  - Centre Jean Perrin, Clermont-Ferrand, Puy-de-Dôme
  - Centre Hospitalier De Pau, Pau, Pyrénées-Atlantiques
  - Institut de Cancerologie Bourgogne, Dijon, Saône-et-Loire
  - CHU Amiens - Picardie Site Sud, Amiens, Somme
  - Institut Gustave Roussy, Villejuif, Val-de-Marne
  - CHI De Fréjus / Saint-Raphael, Fréjus, Var
  - Institut Sainte Catherine, Avignon, Vaucluse
  - CHD Vendee, La Roche-sur-Yon, Vendée
  - Centre Hospitalier Universitaire De Poitiers - Pôle Régional de Cancérologie, Poitiers
  - Institut de Cancérologie de Lorraine, Vandœuvre-lès-Nancy
  - Hopital Tenon, Paris, Île-de-France Region
- Germany (28):
  - Praxisklinik am Rosengarten, Mannheim, Baden-Wurttemberg
  - Universitätsmedizin Mannheim (UMM), Mannheim, Baden-Wurttemberg
  - Hämatologie-Onkologie Zentrum MVZ, Augsburg, Bavaria
  - Universitätsklinikum Augsburg, Augsburg, Bavaria
  - Studienzentrale für das MVZ e.K, Eggenfelden, Bavaria
  - Universitaetsklinikum Erlangen, Erlangen, Bavaria
  - LMU - Klinikum Innenstadt, München, Bavaria
  - Klinikum rechts der Isar, TUM München, München, Bavaria
  - Caritas-Krankenhaus St. Josef - Frauenheilkunde und Geburtshilfe, Regensburg, Bavaria
  - Immanuel Klinik Rüdersdorf, Rüdersdorf, Brandenburg
  - 'Klinikum Esslingen GmbH, Esslingen am Neckar, Esslingen a.N.
  - 'Schwerpunktpraxis Fuer Gynaekologie und Onkologie, Brandenburg, Fuerstenwalde /Spree
  - Klinikum Frankfurt Höchst GmbH, Frankfurt am Main, Hesse
  - Marienhospital Bottrop gGmbH, Bottrop, North Rhine-Westphalia
  - GynOnco Duesseldorf, Düsseldorf, North Rhine-Westphalia
  - Evang. Kliniken Essen-Mitte, Essen, North Rhine-Westphalia
  - Evangelisches Krankenhaus Bethesda, Mönchengladbach, North Rhine-Westphalia
  - Marien Hospital Witten, Witten, North Rhine-Westphalia
  - Klinikum Worms gGmbH, Worms, Rhineland-Palatinate
  - Universitätsklinikum des Saarlandes, Homburg/Saar, Saarland
  - Gemeinschaftspraxis Haematologie - Onkologie, Dresden, Saxony
  - University Hospital Of Leipzig - Frauen- und Kindermedizin, Leipzig, Saxony
  - Universitätsklinikum Schleswig-Holstein, Campus Lübeck, Lübeck, Schleswig-Holstein
  - Praxisklinik Krebsheilkunde, Berlin
  - Helios Klinikum Berlin-Buch, Berlin
  - Charite-Universitaetsmedizin Berlin - Campus Charite Mitte (CCM), Berlin
  - Staedtisches Klinikum Dessau, Dessau
  - Mammazentrum Hamburg MVZ GbR, Hamburg
- Hong Kong (4):
  - Hong Kong Sanatorium & Hospital (HKSH), Happy Valley
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong
  - Queen Mary Hospital - Clinical Oncology, Hong Kong
  - Prince of Wales Hospital (PWH) - The Chinese University of Hong Kong (CUHK) - Clinical Oncology, Shatin
- Hungary (7):
  - University Of Pécs - Oncology dept., Pécs, Baranya
  - Békés Megyei Központi Kórház Pándy Kálmán Tagkórház - Oncology, Gyula, Bekes County
  - Bacs-Kiskun Varmegyei Oktatakorhaz, Kecskemét, Bács-Kiskun county
  - Debreceni Egyetem Klinikai Kozpont, Debrecen, Hajdú-Bihar
  - Nograd Varmegyei Szent Lazar Korhaz, Salgótarján, Szabolcs-Szatmár-Bereg
  - Zala Vármegyei Szent Rafael Korhaz - Onkologiai Osztaly, Zalaegerszeg, Zala County
  - Budapesti Uzsoki Utcai Korhaz, Budapest
- Italy (39):
  - Ospedale Casa Sollievo della Sofferen IRCCS, Opera di San Pio da Pietrelcina, San Giovanni Rotondo, Apulia
  - AOU Cagliari, Monserrato, Cagliari
  - Ist.Oncologico del Mediterraneo, Viagrande, Catania
  - SSD Oncologia Medica Zamagni, IRCCS Azienda Ospedaliero- Universitaria di Bologna, Policlinico di Sant'Orsola, Bologna, Emilia-Romagna
  - IRST Dino Amadori IRCCS, Meldola, Forli-Cesena
  - IRCCS San Gerardo dei Tintori, Monza, Monza E Brianza
  - Azienda Sanitaria Locale Napoli 2 Nord, Frattamaggiore, Napoli
  - Centro di Riferimento Oncologico, IRCCS, Aviano, Pordenone
  - Fond. Piemonte per l'Oncologia - Istituto di Candiolo IRCCS, Candiolo, Torino
  - Divisione di Oncologia Medica ASST Spedali Civili di Brescia, Brescia
  - Ospedale di Cremona, ASST Cremona, Cremona
  - SOD Radioterapia Oncologica, AOU Careggi, Florence
  - Ospedale San Martino IRCCS, Genova
  - Azienda Unità Sanitaria Locale Toscana Nord Ovest, Livorno
  - Ospedale Generale Provinciale di Macerata, Macerata
  - Istituto Nazionale dei Tumori,IRCCS, Milan
  - Istituto Europeo di Oncologia IRCCS, Milan
  - S. C. Oncologia, Centro Oncologico Modenese (COM) - A.O.U. di Modena -Policlinico di Modena, Modena
  - Azienda Ospedaliera Universitaria Federico II, Napoli
  - IRCCS Istituto Nazionale Tumori Fondazione Pascale, Napoli
  - UOC Oncologia - A.O.R.N. "A. Cardarelli", Napoli
  - AOU Maggiore della Carità - Oncologia, Novara
  - Istituto Oncologico Veneto, Padua
  - IRCCS ICS Maugeri, Pavia
  - IRCCS Policlinico San Matteo, Università degli studi di Pavia, Pavia
  - Ospedale Santa Maria Della Misericordia, Perugia
  - PO S.Chiara, AOU Pisana, Pisa
  - PO S Carlo, Azienda Ospedaliera Regionale San Carlo - Oncologia, Potenza
  - Azienda USL Toscana Centro, Prato
  - Azienda Unita Sanitaria Locale della Romagna, Rimini
  - Irccs Crob, Rionero in Vulture
  - Fondazione PU Campus Biomedico, Roma
  - U.O. Ginecologia Oncologica - Fondazione Policlinico A. Gemelli, Roma
  - IRCCS Istituto Nazionale Tumori Regina Elena,UOSD Sperimentazioni di fase IV, Roma
  - AOCO S. Giovanni - Addolorata, Roma
  - Azienda Ospedaliero Universitaria Di Sassari, Sassari
  - Azienda Ospedaliera Universitaria Senese, Siena
  - SOC Oncologia - P.O. "Santa Maria della Misericordia", Udine
  - Ospedale Sacro cuore Don Calabria- Negrar di Valpolicella, Verona
- Malaysia (12):
  - Universiti Sains Malaysia /ID# 200101, Kota Bharu, Kelantan
  - Pantai Hospital Kuala Lumpur, Kuala Lumpur, Kuala Lumpur
  - UKM Medical Centre, Kuala Lumpur, Kuala Lumpur
  - Beacon Hospital, Kuala Lumpur, Kuala Lumpur
  - Universiti Malaya Medical Centre, Kuala Lumpur, Kuala Lumpur
  - Institut Kanser Negara, Putrajaya, Kuala Lumpur
  - Hospital Raja Permaisuri Bainun, Ipoh, Perak
  - Hospital Pulau Pinang - Rheumatology, George Town, Pulau Pinang
  - Institut Perubatan & Pergigian Termaju (IPPT) - USM (Kepala Batas, Pulau Pinang), Kepala Batas, Pulau Pinang
  - Hospital Sultan Ismail, Johor Bahru
  - Hospital Kuala Lumpur, Kuala Lumpur
  - Mahkota Medical Center, Malacca
- Netherlands (4):
  - Elisabeth-TweeSteden Ziekenhuis, Tilburg, North Brabant
  - Albert Schweitzer Ziekenhuis Locatie Dordwijk, Dordrecht, South Holland
  - Haga Ziekenhuis - Internal Medicine, The Hague, South Holland
  - Catharina Ziekenhuis, Eindhoven
- Poland (8):
  - Pratia Poznan, Poznan, Greater Poland Voivodeship
  - Wielkopolskie Centrum Onkologii Oddzial Onkologii Klinicznej i Immunoonkologii, Poznan, Greater Poland Voivodeship
  - Dolnoslaskie Centrum Onkologii, Pulmonologii i Hematologii - Oddzial Onkologii Klinicznej/Chemioterapii, Wroclaw, Lower Silesian Voivodeship
  - Centrum Onkologii Ziemi Lubelskiej im. sw. Jana z Dukli - I Oddzial Onkologii Klinicznej, Lublin, Lubusz Voivodeship
  - Europejskie Centrum Zdrowia Otwock, Szpital im. F. Chopina - Oddział Onkologii Klinicznej, Otwock, Masovian Voivodeship
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie Panstwowy Instytut Badawczy, Warsaw, Masovian Voivodeship
  - Szpitale Pomorskie Sp. z o.o. Oddzial Onkologii Klinicznej, Gdynia, Pomeranian Voivodeship
  - IP Clinic Sp. z o.o., Lodz, Łódź Voivodeship
- Portugal (13):
  - Hospital Beatriz Ângelo. Hospital de Loures - Oncologia Medica, Loures, Lisbon District
  - Hospital De Vila Franca De Xira E.P.E., Vila Franca de Xira, Lisbon District
  - IPO Porto FG, EPE, Porto, Madeira
  - C.H. de Vila Nova de Gaia/Espinho - Oftalmologia, Vila Nova de Gaia, Porto District
  - CHUC - Centro Hospitalar e Universitário de Coimbra, Coimbra
  - Unidade Local de Saúde do Algarve, E. P. E., Faro
  - Instituto Portugues de Oncologia de Lisboa Francisco Gentil - Oncologia Medica, Lisbon
  - ULS Lisboa Ocidental (ULSLO), Lisbon
  - Hospital CUF Descobertas, Lisbon
  - Unidade Local De Saude De Santo Antonio E.P.E., Porto
  - Hospital da Luz de Setubal, Setúbal
  - Unidade Local de Saúde de Arrábida, Setúbal
  - Centro Hospitalar de Trás-os-Montes e Alto Douro, EPE, Vila Real
- Romania (10):
  - Institutul Oncologic Prof Dr Ion Chiricuta Cluj-Napoca, Cluj-Napoca, Cluj
  - Oncolab - Medical Oncology, Craiova, Dolj
  - Onco Clinic Consult - Ambulatory, Craiova, Dolj
  - Centrul de Oncologie Sf. Nectarie, Craiova, Dolj
  - Oncomed - Medical Oncology, Timișoara, Timiș County
  - Spitalul Clinic Filantropia, Bucharest
  - Spitalul Clinic CF Nr 2 Bucuresti, Bucharest
  - Memorial Healthcare International, Bucharest
  - Radiotherapy Center Cluj, Floreşti
  - Institutul Regional de Oncologie Iasi - Medical Oncology, Iași
- Singapore (4):
  - National University Hospital, Singapore, Central Singapore
  - OncoCare Cancer Centre, Singapore, North East
  - Raffles Hospital, Singapore
  - Curie Oncology (Farrer), Singapore
- South Korea (15):
  - Chungbuk National University Hospital, Cheongju-si, Chungcheongbugdo [Ch'ungch'ongbuk-do]
  - CHA Bundang Medical Center, CHA University, Seongnam-si, Gyeonggido
  - Gachon University Gil Medical Center, Incheon, Incheon Gwang'yeogsi [Inch'n-Kwangyokshi]
  - Severance Hospital, Yonsei University Health System, Seoul, Seoul Teugbyeolsi [Seoul-T'ukpyolshi]
  - Asan Medical Center, Seoul, Seoul Teugbyeolsi [Seoul-T'ukpyolshi]
  - Gangnam Severance Hospital - Oncology, Seoul, Seoul Teugbyeolsi [Seoul-T'ukpyolshi]
  - Korea University Guro Hospital, Seoul, Seoul Teugbyeolsi [Seoul-T'ukpyolshi]
  - Korea University Anam Hospital, Seoul, Seoul Teugbyeolsi [Seoul-T'ukpyolshi]
  - Ewha Womans University Mokdong Hospital, Seoul, Seoul Teugbyeolsi [Seoul-T'ukpyolshi]
  - Inje University Haeundae Paik Hospital, Busan
  - National Cancer Center, Gyeonggi-do
  - Ajou University Hospital, Gyeonggi-do
  - Seoul National University Hospital, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
  - Ulsan University Hospital, Ulsan
- Spain (33):
  - Hospital Alvaro Cunqueiro, Vigo, A Coruña
  - Hospital Universitario Virgen del Rocío, Seville, Andalusia
  - H. Virgen de Valme, Seville, Andalusia
  - ICO Badalona-Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitari General de Catalunya, Sant Cugat del Vallès, Barcelona
  - Hospital de Sant Joan Despi Moises Broggi, Sant Joan Despí, Barcelona
  - Hospital Universitario de Canarias, San Cristóbal de La Laguna, Canary Islands
  - Hospital Universitario Rey Juan Carlos, Móstoles, Madrid
  - Hospital Clínico Universitario Virgen De La Arrixaca, El Palmar, Murcia
  - Fundación Instituto Valenciano Oncologia, Valencia, Navarre
  - Complexo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital Clinic De Barcelona - Oncología Médica, Barcelona
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario de Jaén, Jaén
  - H.U. Insular Gran Canaria, Las Palmas de Gran Canaria
  - H.U Arnau De Vilanova Lleida, Lleida
  - Hospital Universitario Lucus Augusti, Lugo
  - Hospital Beata Maria Ana, Madrid
  - Hospital General Universitario Gregorio Marañón - Oncology, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen De La Victoria, Málaga
  - Hospital Regional Universitario de Málaga (Hospital Civil), Málaga
  - Hospital Universitario de Santiago, Santiago de Compostela
  - Hospital Universitario Virgen de la Macarena - Oncología Médica, Seville
  - Hospital Clinico Universitario De Valencia, Valencia
  - Hospital Quironsalud Valencia, Valencia
  - Hospital Clínico Universitario Lozano Blesa - Oncología Médica, Zaragoza
- Switzerland (12):
  - Tumor Zentrum Aarau, Aarau, Aargau (de)
  - Kantonsspital Badenv, Baden, Aargau (de)
  - Kantonsspital Baselland, Liestal, Basel-Landschaft (de)
  - Universitätsspital Basel, Basel, Basel-Stadt (de)
  - HOCH Health Ostschweiz - Kantonsspital St.Gallen, Sankt Gallen, Sankt Gallen (de)
  - Centre Hospitalier Universitaire Vaudois (CHUV)Département d'oncologie, Lausanne, Vaud (fr)
  - Kantonsspital Winterthur, Winterthur, Zürich (de)
  - Brust-Zentrum AG Zurich, Zurich, Zürich (de)
  - Inselspital, Universitätsspital Bern, Bern
  - Hopitaux Universitaires de Geneve (HUG) - Hopital Cantonal, Geneva
  - Spitaeler Schaffhausen Kantonspital, Schaffhausen
  - Universitätsspital Zürich, Zurich
- Taiwan (12):
  - Kuang Tien General Hospital - Shalu Xiangshang Division - Hemato-Oncology, Taichung, Taichung
  - Taipei Tzu Chi Hospital, Buddhist Tzu Chi Medical Foundation, New Taipei City, Taipei
  - Taipei Medical University - Shuang Ho Hospital Ministry of Health and Welfare - Hematology & Oncology, New Taipei City, Taipei
  - Taipei Veterans General Hospital - Hematology, Taipei City, Taipei
  - National Defense Medical Center (NDMC) - Tri-Service General Hospital - Neihu Branch, Taipei City, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center - Hematology, Taipei, Taoyuan
  - Chang Gung Medical Foundation - LinKou Chang Gung Memorial Hospital - Breast Surgery, Taiyuan, Taoyuan
  - Changhua Christian Medical Foundation Changhua Christian Hospital, Changhua
  - China Medical University Hospital - Breast Surgery, Taichung
  - National Cheng Kung University Hospital, Tainan
  - Chi Mei Medical Center - Liouying - Oncology, Tainan
  - National Taiwan University Hospital - Surgery, Taipei
- Turkey (Türkiye) (26):
  - Baskent Universitesi Adana Uygulama ve Arastirma Merkezi, Adana, Adana/ Yuregir
  - Sakarya Egit ve Aras Hast, Sakarya, Adapazari
  - Dr Abdurrahman Yurtaslan EAH, Ankara, Ankara/ Yenimahalle
  - Memorial Ankara Hastanesi, Ankara, Ankara/Cankaya
  - Ankara City Hospital - Medical Oncology, Ankara, Cankaya/Ankara
  - Prof. Dr. Suleyman Yalcin Sehir Hastanesi, Kadıköy, Istanbul
  - VM MedicalPark Pendik Hospital, Istanbul, Istanbul/Pendik
  - Dokuz Eylul Universitesi - Tip Fakultesi, Balçova, İzmir
  - Kocaeli Uni Egt ve Uyg Hast, İzmit, Kocaeli
  - Necmettin Erbakan Universitesi Tip Fakultesi Hastanesi, Konya, Meram/Konya
  - VM Medical Park Mersin Hastanesi, Mersin, Mersin/Mezitli
  - Acibadem Maslak Hospital, Istanbul, Samsun
  - Acibadem Atasehir Hospital, Istanbul, Samsun
  - Medical Park Seyhan Hospital, Adana, Seyhan/Adana
  - Gazi Uni Hast, Ankara, Yenimahalle/Ankara
  - Adana Sehir Egitim ve Arastirma Hastanesi, Adana, Yüregir
  - Ankara Etlik Sehir Hastanesi - Tıbbi Onkoloji, Ankara
  - Hacettepe University Medical Faculty - Medical Oncology, Ankara
  - Gulhane Training and Research Hospital, Ankara
  - Ankara Universitesi Tip Fakultesi Cebeci Arastirma Ve Uygulama Hastanesi, Ankara
  - Adnan Menderes Universitesi - Uygulama ve Arastirma Hastanesi, Aydin
  - Dicle Universitesi Hastanesi, Diyarbakır
  - Medical Park Florya Hastanesi, Istanbul
  - Acibadem Altunizade Hospital, Istanbul
  - Medical Point Izmir Hospital, Izmir
  - VM Medical Park Samsun Hospital - Medical oncology, Samsun
- United Kingdom (13):
  - Royal Cornwall Hospital (RCH) - Sunrise Centre, Truro, Cornwall
  - Whittington Health NHS Trust - Whittington Hospital, London, England
  - Cheltenham General Hospital, Cheltenham, Gloucestershire
  - Mount Vernon Cancer Centre - Main Site, Northwood, Greater London
  - Blackpool Victoria Hospital, Blackpool, Lancashire
  - Royal Preston Hospital, Preston, Lancashire
  - University College London Hospitals, London, London, City of
  - St John's Hospital - NHS Lothian, Livingston, Scotland
  - Musgrove Park Hospital, Taunton, Somerset
  - Western General Hospital, Edinburgh
  - Leeds Cancer Centre, Leeds
  - St Bartholomew's Hospital, London
  - Maidstone Hospital Kent Oncology Centre, Maidstone